CLINICAL TRIAL: NCT06584214
Title: A Prospective, Multi-centre Study to Evaluate the Diagnostic Sensitivity and Specificity of the Determine™ Syphilis Advanced Test.
Brief Title: Evaluation of the Diagnostic Sensitivity and Specificity of the Determine™ Syphilis Advanced Test.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Rapid Dx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D10159847 (7D34VAL24-002)
Record Dates: First submitted 2024-08-29; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Syphilis Infection

STUDY DESIGN:
Masking Description: Study staff performing the testing using the Determine™ Syphilis Advanced and Determine™ Syphilis TP testing will be blinded to the participants' syphilis infection status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic test: Determine™ Syphilis Advanced test (Experimental): Diagnostic test: Testing using the Determine™ Syphilis Advanced test will be conducted by study staff members.
  Interventions: Diagnostic Test: Diagnostic test: Determine™ Syphilis Advanced test

INTERVENTIONS:
Diagnostic Test: Diagnostic test: Determine™ Syphilis Advanced test — The Determine™ Syphilis Advanced test is intended as an aid in detecting antibodies to Treponema pallidum in individuals with current or past infection.

SUMMARY:
This is a prospective, multi-centre study which will evaluate the diagnostic sensitivity and specificity of the Determine™ Syphilis Advanced test. The test is intended for professional use and the performance evaluation will be performed by professional healthcare and laboratory staff. The study will also have a retrospective study arm. The Determine™ Syphilis Advanced validation will be conducted in accordance with the World Health Organization's TSS-6 guidance on Syphilis rapid diagnostic tests, ISO 20916 (In vitro diagnostic medical devices - Clinical performance studies using specimens from human subjects - Good study practice), the study protocol, Good Clinical Practice and the respective local medical device laws.

DETAILED DESCRIPTION:
Syphilis is a sexually transmitted infection (STI) caused by the spirochete Treponema pallidum subspecies. Globally, there were an estimated 7.1 million adults between 15 and 49 years of age who acquired syphilis in 2020. Syphilis is transmitted through sexual contact with infectious lesions, through blood transfusions and from mother-to-child during pregnancy; most infections are asymptomatic or unrecognized. Without treatment, the disease lasts for many years and is divided into stages: primary syphilis, secondary syphilis and latent syphilis. Mother-to-child transmission of syphilis (congenital syphilis) can adversely affect the foetus, but this can be averted by early detection and treatment of the mother during pregnancy.

Determine™ Syphilis Advanced is an in vitro, visually read, qualitative immunoassay for the detection of antibodies to Treponema pallidum, in human capillary and venous whole blood, plasma or serum.

The test is intended for professional use, and the performance evaluation will be performed by professional healthcare and laboratory staff. Results for all sample types (capillary and venous whole blood, plasma or serum) will be evaluated against reference test results. In addition, for a sub-cohort, the Determine™ Syphilis Advanced test will be compared with the commercially available Determine™ Syphilis TP and the SERODIA-TPPA tests. Study staff performing the testing using the Determine™ Syphilis Advanced will be blinded to the participants' syphilis infection status and all other study syphilis test results. The study will enrol prospective participants, and will also have a retrospective study group.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older.
* The participant has confirmed previous / current syphilis according to their medical history, or the participant has unknown or negative syphilis infection status.
* The participant agrees to provide written informed consent.
* The participant agrees to complete all aspects of the study.

Additional inclusion criteria for frozen samples:

* The ethics committee-required written informed consent for study testing, or required documentation for sample use from a commercial vendor, is available.
* Sufficient volume for testing is available and the sample quality is adequate (for example no significant sample hemolysis)
* The sample must have been collected in EDTA vacutainers or serum tubes, processed to plasma and the plasma frozen within 36 hours of blood collection.

Exclusion Criteria:

* Participant has already participated in this study on a previous occasion.
* Participant is deemed vulnerable and / or unfit for participation in the study by the Investigator.
* Participant is unwilling or unable to provide informed consent.
* Participant is currently enrolled in a study to evaluate an investigational new drug or vaccine.

Additional exclusion criteria for frozen samples

* The sample has undergone more than one freeze thaw cycle
* The sample has been kept at -20 °C (± 5 °C) longer than 12 months. If the sample has been kept longer than 12 months, the storage temperature must have been colder than -20 °C (± 5 °C).

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To determine the diagnostic sensitivity and specificity of the Determine™ Syphilis Advanced test results using fingerstick capillary whole blood, venous whole blood, serum and venous plasma, when the test is performed by professional users. | 4 months
  The diagnostic sensitivity and specificity of the Determine™ Syphilis Advanced test will be evaluated versus laboratory reference testing.
To compare the performance of the Determine™ Syphilis Advanced test with two commercially available similar tests | 4 months
  The Determine™ Syphilis Advanced test will be compared with two commercially available tests. These tests are the TPPA test (SERODIA-TPPA, Fujirebio) and the Determine™ Syphilis TP (Abbott) test.

SECONDARY OUTCOMES:
To evaluate the usability through completion of a user experience questionnaire. | 4 months
  A user experience questionnaire will be completed by study healthcare staff. The users will evaluate the ease of use, and confidence in correct performance, of various test steps and result interpretation. The response options are ranked on a scale of 1-5. where option 1 stands for Very easy, or Very confident as applicable, and 5 stands for Very Difficult, or Very unsure as applicable.
To determine the stability of venous whole blood, serum and plasma samples for use with Determine™ Syphilis Advanced, after refrigeration . | 4 months
  Venous whole blood, serum and plasma will be stored at 2-8 degrees Celsius during 7 days before testing with Determine™ Syphilis Advanced.

CONTACTS AND LOCATIONS:
Overall Officials: Pontiano Kaleebu, Professor, MD PhD, Principal Investigator — MRC/UVRI and LSHTM Uganda Research Unit
Locations (1):
- Uganda Virus Research Institute, Entebbe, Uganda

IPD SHARING:
Plan to Share IPD: No